CLINICAL TRIAL: NCT00100633
Title: Immunologic Effects of CpG ODN Administration to HIV Uninfected and HIV Infected Patients
Brief Title: Safety of and Immune Response to a Hepatitis B Virus Vaccine Given With a Booster (CpG7909 ODN) in HIV Infected and HIV Uninfected People
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Michael M. Lederman/Professor of Medicine, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01AI055793 (NIH); P01AI055793 (NIH)
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections; Hepatitis B
Keywords: Hepatitis B Vaccine; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Drug: CpG7909 oligodeoxynucleotides (ODN)
Biological: Hepatitis B virus vaccine

SUMMARY:
The purpose of the study is to determine the safety of and immune response to a hepatitis B virus vaccine series given with a boosting agent, CpG7909 oligodeoxynucleotides (ODN), in HIV infected and HIV uninfected individuals who previously failed to develop a response to hepatitis B vaccine.

Study hypothesis: Administration of CpG7909 ODN together with recombinant hepatitis B vaccine will result in increased frequency and magnitude of response to vaccine in individuals who have previously failed to mount a response to vaccination, and that in HIV infected subjects with detectable plasma viremia, it will lead to the enhancement of HIV-specific responses.

DETAILED DESCRIPTION:
As HIV disease progresses in HIV infected people, their immune responses to infectious and other foreign invaders becomes weaker; in particular, the cellular (T-cell) immune response is particularly affected by HIV. A boosting agent called CpG7909 ODN may be an ideal adjuvant for vaccines given to HIV infected people, because it may help elicit an increased CD8 T-cell response. This study will evaluate the safety of and immune response to a hepatitis B virus vaccine series given with CpG7909 ODN in HIV infected and uninfected people.

There will be three groups in this study; participants will be stratified by baseline CD4 counts and viral load. Within each group, participants will be randomly assigned to receive 3 injections of hepatitis B vaccine with CpG7909 ODN or 3 injections of hepatitis B vaccine alone. Injections will be given at study entry and Months 1 and 6. There will be 10 study visits; a physical exam and blood collection will occur at each visit.

ELIGIBILITY:
Inclusion Criteria for HIV Infected Participants:

* HIV-1 infection
* If receiving combination antiretroviral therapy (ART), must have been on ART for at least 3 months prior to study entry. Patients who anticipate a change in treatment (either initiating ART or stopping ART) in the next 7 months are not eligible.
* CD4 count of 250 cells/mm3 or greater
* Negative HBsAb, HBsAg, and HBcAb
* Willing to use acceptable forms of contraception while on study treatment and for 24 weeks after study treatment has ended

Inclusion Criteria for HIV Uninfected Participants:

* HIV uninfected
* Negative HBsAb, HBsAg, and HBcAb
* Willing to use acceptable forms of contraception while on study treatment and for 24 weeks after study treatment has ended

Exclusion Criteria for All Participants:

* Cancer. Participants with squamous cell or basal cell skin cancer are not excluded.
* Autoimmune disease
* Immunosuppressive medications. People who use or have used corticosteroid nasal sprays are not excluded. People who have received fewer than 2 weeks of systemic corticosteroids with the last dose over a month prior to study entry are not excluded.
* Any medical or psychiatric condition or occupational responsibilities that may interfere with the study
* Immunomodulator or investigational agent therapy within 30 days prior to study entry
* Allergy/sensitivity to study drugs or their formulations, including thimerosal
* Current drug or alcohol use that, in the opinion of the investigator, would interfere with the study
* Active hepatitis C virus infection, as indicated by serum antibodies to HCV AND detectable HCV RNA in plasma
* Blood clotting abnormalities
* Any other condition that, in the opinion of the investigator, might interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-12; Primary Completion 2007-02 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of HIV peptides to which HIV infected patients respond using ELISPOT (CpG vs. no CpG in HIV infected participants)
total number of CD8+ lymphocytes responding after HIV-peptide stimulation using ELISPOT (CpG vs. no CpG in HIV infected participants)
safety

SECONDARY OUTCOMES:
Percentage of patients who develop protective hepatitis B (HB) antibody concentration (CpG vs. no CpG in HIV infected participants)
percentage of patients who develop HB specific CD8+ lymphocyte responses using ELISPOT (CpG vs. no CpG in HIV infected participants)
percentage of patients who develop HB specific CD8+ lymphocyte responses using ELISPOT (CpG vs. no CpG in all participants)
percentage of patients who develop CD8+ lymphocyte proliferative responses as measured using CFSE (CpG vs. no CpG in HIV infected participants)
percentage of patients who develop CD8+ lymphocyte proliferative responses as measured using CFSE (CpG vs. no CpG in all participants)
expression of costimulatory molecules on B-cells in peripheral blood (CpG vs. no CpG in HIV infected participants)
expression of costimulatory molecules on B-cells in peripheral blood (CpG recipients, HIV infected vs. uninfected participants)
spontaneous IFN-gamma production in peripheral blood (CpG recipients, HIV infected vs. uninfected participants)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Lederman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Background] Jiang JQ, Patrick A, Moss RB, Rosenthal KL. CD8+ T-cell-mediated cross-clade protection in the genital tract following intranasal immunization with inactivated human immunodeficiency virus antigen plus CpG oligodeoxynucleotides. J Virol. 2005 Jan;79(1):393-400. doi: 10.1128/JVI.79.1.393-400.2005. PMID 15596832
- [Background] Schlaepfer E, Audige A, von Beust B, Manolova V, Weber M, Joller H, Bachmann MF, Kundig TM, Speck RF. CpG oligodeoxynucleotides block human immunodeficiency virus type 1 replication in human lymphoid tissue infected ex vivo. J Virol. 2004 Nov;78(22):12344-54. doi: 10.1128/JVI.78.22.12344-12354.2004. PMID 15507621